CLINICAL TRIAL: NCT04012580
Title: Examining The Acceptability and Effectiveness of Transdiagnostic, Internet-Delivered Cognitive Behaviour Therapy for Symptoms of Postpartum Anxiety and Depression: A Randomized Controlled Trial
Brief Title: Examining the Effectiveness of Transdiagnostic, Internet-Delivered Cognitive Behaviour Therapy in New Mothers Experiencing Anxiety and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-077
Record Dates: First submitted 2019-07-04; First posted 2019-07-09 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2020-11

CONDITIONS: Depression, Postpartum; Anxiety
Keywords: postpartum; depression; anxiety; internet-delivered cognitive behaviour therapy; randomized controlled trial; therapist-assistance
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapist-assisted ICBT (Experimental): An 8-week transdiagnostic internet-delivered cognitive behavioural therapy (ICBT) will be delivered to participants. In addition to the program, participants will receive support from registered social workers, psychologists or supervised graduate students, with experience delivering ICBT, with contact provided on a weekly basis.
  Interventions: Behavioral: Therapist-assisted ICBT
- Treatment as usual control (No Intervention): Participants will not receive access to the transdiagnostic internet-delivered cognitive behavioural therapy (ICBT) program for 12-weeks. Participants will be permitted to access community resources (e.g., support groups). After 12-weeks, participants will be offered the program although their treatment data will not be included in the current study.

INTERVENTIONS:
Behavioral: Therapist-assisted ICBT — An 8-week transdiagnostic internet-delivered cognitive behavioural therapy (ICBT) will be delivered to participants. In addition to the online program, therapists, registered social workers, psychologists or supervised graduate students will provide support by email once a week.
  Arms: Therapist-assisted ICBT

SUMMARY:
In the proposed study, the investigators will examine the efficacy of transdiagnostic, Internet-delivered cognitive behaviour therapy (ICBT) in the treatment of postpartum anxiety and depression. Half of participants will receive the treatment immediately, and half of the participants will be assigned to a treatment-as-usual control condition. Participants assigned to the control condition will be offered the treatment after a 12-week waiting period, although data from this portion will not be included in the current study. All participants will complete questionnaires prior to the start of the treatment, following treatment (or corresponding 8-week waiting period), at 1-months follow-up (or corresponding 12-week waiting period), and at 6-months follow-up (in those assigned to the treatment condition). Further, those who receive the treatment will complete questionnaires on a weekly basis. The primary outcome measures include anxiety and depression. As part of the battery of questionnaires administered after the completion of the program, participants will be asked to rate the program content, the overall service, and their satisfaction with the program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* female
* have given birth and have a child under one year of age
* score of 10 or above on EPDS or a score of 9 or above on the GAD-7
* be a resident of Saskatchewan
* have access to a secure computer and the Internet, and be comfortable using technology
* be available to work through treatment each week
* be willing to provide a medical contact as an emergency contact

Exclusion Criteria:

* younger than 18 years
* not female
* have not given birth to a child less than one year of age
* are experiencing minimal to no symptoms of anxiety and/or depression
* are not a resident of Saskatchewan
* have been hospitalized within the last year for mental health and/or suicide risk concerns;
* have unmanaged problems with alcohol, drugs, psychosis or mania, or are at increased suicide risk (specific plans and intent reflected by the Suicide Behaviors Questionnaire-Revised)
* started a new psychotropic medication within the past month
* do not have access to a secure computer and the Internet or is not comfortable using technology
* are not available to work through treatment each week
* are not willing to provide a medical contact as an emergency contact

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Change in postpartum depression | Baseline, weeks 1-9, 13, and 37
  Measured by the Edinburgh Postnatal Depression Scale (EPDS). 10 items are summed into a total score ranging from 0 to 30, with higher scores indicating more severe depression.
Change in anxiety | Baseline, weeks 1-9, 13, and 37
  Measured by the Generalized Anxiety Disorder Scale 7-Item (GAD-7). 7 items are summed into a total score ranging from 0 to 21, with higher scores indicating more severe self-reported levels of anxiety.

SECONDARY OUTCOMES:
Change in depression | Baseline, weeks 1-9, 13, and 37
  Measured by the Patient Health Questionnaire 9-Item (PHQ-9). 9 items are summed into a total score, with scores ranging from 0 to 27. Higher scores are associated with higher depression severity.
Change in depression, anxiety, stress | Baseline, 8 weeks, 1 month, and 6 months
  Measured by the Depression and Anxiety Stress Scales (DASS-21). 21 items are summed into a total score ranging from 0 to 42, with higher scores indicating more severe symptoms with respect to the depression, anxiety, and stress subscales.
Mother-infant bonding | Baseline, weeks 9, 13, and 37
  Measured by the Postnatal Bonding Questionnaire (PBQ). 25 items are summed into a total score ranging from 0 to 125, with higher scores indicating more reported difficulties bonding with one's baby.
Relationship satisfaction | Baseline, weeks 9, 13, and 37
  Measured by the Dyadic Adjustment Scale-7 item (DAS-7). 7 items are summed into a total score ranging from 0 to 32, with higher scores indicating greater perceived relationship quality.
Treatment credibility | Baseline and week 9
  Measured by the Credibility/Expectancy Questionnaire (CEQ). 6 items are summed into a total score and two subscales (credibility and expectancy). Total scores can range from 3 to 27, with higher scores representing greater perceptions of ICBT credibility.
Therapeutic alliance | 9 weeks following baseline
  Measured by the Working Alliance Inventory-Short Revised (WAI-SR). Scores are summed into three sub-total scores, which respectively assess various domains of the therapeutic relationship (i.e., goal, task, and bond). Sub-total scores each range between 5 and 20, with higher scores representing better therapeutic relationship in each of the three domains assessed.
Treatment satisfaction | 9 weeks following baseline
  Measured by the Treatment Satisfaction Questionnaire (TSQ). 6 items are scored using various scales. Descriptive statistics are produced for each item.
Adverse effects | 9 weeks following baseline
  Measured by questions assessing whether participants encountered any adverse effects of treatment, developed any new psychological symptoms, or experienced any unexpected events over the course of treatment
Service utilization | Weeks 9, 13, and 37
  Measured by a series of questions asking participants whether they accessed additional services or support

CONTACTS AND LOCATIONS:
Overall Officials: Marcie Nugent, MSW, Study Director — University of Regina
Locations (1):
- Online Therapy Unit, University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suchan V, Peynenburg V, Thiessen D, Nugent M, Dear B, Titov N, Hadjistavropoulos H. Transdiagnostic Internet-Delivered Cognitive Behavioral Therapy for Symptoms of Postpartum Anxiety and Depression: Feasibility Randomized Controlled Trial. JMIR Form Res. 2022 Sep 6;6(9):e37216. doi: 10.2196/37216. PMID 36066958